CLINICAL TRIAL: NCT01388725
Title: Comparison of the Value of Serum sTREM-1, sCD163, PCT, CRP Concentrations, WBC Count and SOFA Score During Sepsis and Their Clinical Informative Value in Predicting Outcome
Brief Title: Comparison the Value of Several Biomarkers of Sepsis
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Lixin Xie, Department Of Respiratory Diseases, Chinese PLA General Hospital
Other Study IDs: 20090923-001,20100701-002; 2009BAI86B03 (Other Grant/Funding Number: Chinese National Science & Technology Pillar Program)
Record Dates: First submitted 2011-07-05; First posted 2011-07-07 (Estimated); Last update posted 2011-07-07 (Estimated); Status verified 2010-07

CONDITIONS: Systemic Inflammatory Response Syndrome; Sepsis
Keywords: sTREM-1; sCD163; PCT; CRP; WBC count; SOFA score; SIRS; sepsis; severity; prognosis
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome; Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- SIRS: (1) temperature > 38oC or < 36oC; (2) pulse rate > 90 beats/min; (3) ventilation rate > 20 breaths/min or hyperventilation with a partial pressure of arterial carbon dioxide (PaCO2) < 32 mmHg; (4) white blood cell (WBC) count >1 2,000μL-1 or < 4000 μL-1 , or > 10% immature cells.
- Sepsis: SIRS + infection

SUMMARY:
The purpose of this study is to describe the value of serum sTREM (soluble triggering receptor expressed on myeloid cells)-1, sCD163, procalcitonin (PCT), C-reactive protein (CRP) concentrations, white blood cell (WBC) count and SOFA score during sepsis and their clinical informative value in predicting outcome.

DETAILED DESCRIPTION:
The investigators enrolled 130 subjects admitted to an ICU: 30 cases with systemic inflammatory response syndrome (SIRS), 36 cases with sepsis, 35 cases with and 29 with septic shock. Results for sTREM (soluble triggering receptor expressed on myeloid cells)-1, sCD163, procalcitonin (PCT), C-reactive protein (CRP) concentrations, white blood cell (WBC) count and SOFA score were recorded on days 1, 3, 5, 7, 10, and 14.

ELIGIBILITY:
Inclusion Criteria:

* Male and female aged 18 years old and over;
* Clinically suspected infection;
* Fulfilled at least two criteria of systemic inflammatory response syndrome (a) core temperature higher than 38 °C or lower than 36 °C (b)respiratory rate above 20/min, or PCO2 below 32 mmHg (c) pulse rate above 90/min, and (d) white blood cell count greater than 12,000/μl or lower than < 4,000/μl or less than 10% of bands.

Exclusion Criteria:

* Those who fulfilled one below:
* neutropenia (≤ 500 neutrophils/mm3)
* HIV infection, and
* patients or their relatives refused

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Between September 2009 and July 2011, inpatients were included who were in the intensive care units (ICU) of the Department of Respiratory Disease, the Emergency Department, and the Department of Surgery of the Chinese People's Liberation Army General Hospital.
Sampling Method: Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2009-09; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Patients Outcome | 28 days
  The survival time of patients more than 28 days is defined as survival. The survival time of patients less than 28 days is defined as death

CONTACTS AND LOCATIONS:
Overall Officials: Xie Lixin, Doctor, Study Director — Department Of Respiratory Diseases, Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China